CLINICAL TRIAL: NCT02272426
Title: The Safety and Tolerability of an Aerobic and Resistance Exercise Program With Cognitive Training Post-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: American Heart Association (Other); Bugher Foundation (Unknown)
Responsible Party: Principal Investigator, Sebastian Koch, Professor of Neurology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20140203
Record Dates: First submitted 2014-10-01; First posted 2014-10-23 (Estimated); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Cerebral Stroke
Keywords: Stroke; Exercise Training; Cognitive Training; Quality of Life
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CARET + CTI (Experimental): Combined Aerobic and Resistance Exercise Training (CARET) plus Cognitive Training Intervention (CTI)
  Interventions: Behavioral: CARET; Behavioral: CTI
- Sham CARET + Sham CTI (Sham Comparator): Control group Sham Combined Aerobic and Resistance Exercise Training (CARET) plus Sham Cognitive Training Intervention (CTI)
  Interventions: Behavioral: Sham CARET; Behavioral: Sham CTI

INTERVENTIONS:
Behavioral: CARET — Combined Aerobic and Resistance Exercise Training
  Arms: CARET + CTI
Behavioral: CTI — Cognitive Training Intervention
  Arms: CARET + CTI
Behavioral: Sham CARET — Sham Combined Aerobic and Resistance Exercise Training
  Arms: Sham CARET + Sham CTI
Behavioral: Sham CTI — Sham Cognitive Training Intervention
  Arms: Sham CARET + Sham CTI

SUMMARY:
It is estimated that 2 out of 3 patients with a stroke have some problems with their memory, difficulties performing certain tasks, making decisions and learning new things. In addition, many stroke patients do not get regular exercise and are often sedentary. Both physical and cognitive exercise have the potential to improve quality of life, cognition, and overall health, but the safety and tolerability of such interventions is not clear in stroke patients. The investigators will examine these outcomes by allocating stroke survivor participants to one of two groups: a combined exercise and cognitive training program and a sham control group.

DETAILED DESCRIPTION:
Stroke is well recognized as the leading cause of disability in the United States. Cognitive deficits after stroke are common, even in those without dementia prior to the event, and stroke patients with worse cognition on hospital admission have worse outcomes. Cognitive deficits contribute to stroke-related disability and mortality. Evidence suggests an interaction between cognitive deficits and physical limitations, and cognitive rehabilitation may improve functional outcomes post stroke. Recent data also suggest that both cognitive training and exercise interventions improve cognition in stroke patients, but few randomized trials of these interventions, alone or in combination, have been conducted.

We will study the effects of a Combined Aerobic and Resistance Exercise Training (CARET) program and CTI interventions on the primary outcome of safety, feasibility, and adherence among ischemic or hemorrhagic stroke survivors with mild to moderate disability. We hypothesize that these interventions are safe and tolerable, and that they will lead to improvements in our secondary outcomes of cognitive performance and quality of life. We will also explore the role of Brain Derived Neurotrophic Factor in cognitive changes related to the physical exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic or hemorrhagic stroke
* Modified Rankin Score (mRS) of <4 at screening
* Recently discharged from the hospital or rehabilitation program
* Male or female ≥18 years of age
* Less than ideal physical activity ≥ 3 months prior to enrollment (less than ideal physical (as defined by the American Heart Association)
* Able to walk ≥10 meters with or without assistance

Exclusion Criteria:

* Unable to follow instructions for exercise and cognitive interventions
* Any uncontrolled medical condition expected to limit life expectancy or interfere with participation in the trial (i.e. unstable cancer, severe depression or anxiety by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria)
* Abnormal stress test, as determined by the treating physician (unless cardiology clearance provided)
* Active substance abuse or alcohol dependence
* Less than 6th grade reading level
* Uncorrected vision or hearing deficits that would preclude administration of the cognitive measures
* Unwilling or unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-11; Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent serious adverse events | At 12 weeks visit (post-intervention)
  To assess the number of participants with serious adverse events related to the interventions, comparing active groups versus the sham group.
Adherence to a 12-week combined exercise and cognitive training protocol versus a sham group | At 12 weeks visit (post-intervention)
  To assess participant adherence in the intervention group versus the sham group, comparing time on study.

SECONDARY OUTCOMES:
Change in Cognitive Performance on cognitive neuropsychological battery done at pre, post and 6 month follow-up visits | Baseline to 6 months follow up
  Global cognitive performance will be compared for the intervention groups versus the sham group, using a cognitive assessment battery.
Change in Health Related Quality of Life - Depression | Baseline to 6 months follow up measure.
  As measured by Center for Epidemiologic Studies Depression Scale (CES-D). Minimum score 0, maximum score 60, and a score of 16 or higher indicates clinical depression.
Change in Health Related Quality of Life - Daily Activities | Baseline to 6 months follow up
  As measured by Stroke impact scale scores measuring health related quality of life. Minimum score 16, maximum score 80. Higher scores indicate higher level of functionality in participants, while lower scores indicate a lower level of functionality.
Change in blood plasma concentration of Brain Derived Neurotrophic Factor | Baseline to 6 month follow up
  Brain-derived neurotrophic factor (BDNF) levels will be compared between the exercise group and the sham group at baseline and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Koch, M.D., Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami Hospital, Miami, Florida

REFERENCES:
- [Derived] Koch S, Tiozzo E, Simonetto M, Loewenstein D, Wright CB, Dong C, Bustillo A, Perez-Pinzon M, Dave KR, Gutierrez CM, Lewis JE, Flothmann M, Mendoza-Puccini MC, Junco B, Rodriguez Z, Gomes-Osman J, Rundek T, Sacco RL. Randomized Trial of Combined Aerobic, Resistance, and Cognitive Training to Improve Recovery From Stroke: Feasibility and Safety. J Am Heart Assoc. 2020 May 18;9(10):e015377. doi: 10.1161/JAHA.119.015377. Epub 2020 May 12. PMID 32394777